CLINICAL TRIAL: NCT07148362
Title: Comparison of Upper Extremity Exercise Capacity, Muscle Oxygenation, and Balance in Pediatric Cystic Fibrosis and Primary Ciliary Dyskinesia
Brief Title: Upper Extremity Exercise Capacity, Muscle Oxygenation, and Balance in Pediatric CF and PCD
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof., Gazi University
Other Study IDs: 2025-557
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis (CF); Primary Ciliary Dyskinesia (PCD)
Keywords: cystic fibrosis; primary ciliary dykinesia; balance; muscle oxygenation; exercise tolerance; upper extremity
MeSH Terms: conditions — Cystic Fibrosis; Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Cystic fibrosis: Upper extremity functional exercise capacity was evaluated using the 6-minute pegboard and ring test, pulmonary function using spirometry, peripheral muscle strength using a hand-held dynamometer, muscle oxygenation using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD), static balance using the "Biosway Portable Balance System", and dynamic balance assessment using the Y balance test.
- Patients with Primary ciliary dyskinesia: Upper extremity functional exercise capacity was evaluated using the 6-minute pegboard and ring test, pulmonary function using spirometry, peripheral muscle strength using a hand-held dynamometer, muscle oxygenation using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD), static balance using the "Biosway Portable Balance System", and dynamic balance assessment using the Y balance test.
- Healthy controls: Upper extremity functional exercise capacity was evaluated using the 6-minute pegboard and ring test, pulmonary function using spirometry, peripheral muscle strength using a hand-held dynamometer, muscle oxygenation using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD), static balance using the "Biosway Portable Balance System", and dynamic balance assessment using the Y balance test.

SUMMARY:
The number of studies evaluating respiratory functions and upper extremity functional exercise capacity in patients with CF and PCD is limited in the literature. There are no studies comparing upper extremity functional exercise capacity and upper extremity muscle oxygenation in patients with CF and PCD. The aim of our study is to compare respiratory function, upper extremity functional exercise capacity, peripheral muscle strength, muscle oxygenation, and balance in CF, PCD, and healthy children.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an autosomal recessive, monogenic disorder caused by mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene. In individuals with CF, infections, inflammation, mucus plugging, nutritional deficiencies, pulmonary exacerbations, and respiratory tract diseases contribute to a decline in pulmonary function. Increased airway resistance, air trapping, and reduced airflow rates lead to a decrease in lung capacities. Primary ciliary dyskinesia (PCD) is a genetically heterogeneous disorder caused by the absence or dysfunction of motile cilia. In PCD, pulmonary function is affected from early in life and remains below reference values across all age groups and both sexes. Decreased muscle strength has been demonstrated in both CF and PCD patients. In chronic obstructive pulmonary disease (COPD), pulmonary function and limb muscle strength are important determinants of exercise capacity. There is a limited number of studies in the literature assessing pulmonary function and upper extremity functional exercise capacity in patients with CF and PCD. Furthermore, to our knowledge, no studies have compared upper extremity functional exercise capacity and upper extremity muscle oxygenation between patients with CF and PCD. The aim of this study is to compare pulmonary function, upper extremity functional exercise capacity, peripheral muscle strength, muscle oxygenation, and balance among children with CF, children with PCD, and healthy controls. The study was planned as cross-sectional and retrospective. The patient group will include individuals diagnosed with CF and PCD, aged between 6 and 18 years, receiving standard medical treatment. The healthy group will include individuals aged between 6 and 18 years without any known chronic disease. Individuals' respiratory functions, upper extremity functional exercise capacity, peripheral muscle strength, muscle oxygenation, and balance will be evaluated. Upper extremity functional exercise capacity was evaluated using the 6-minute pegboard and ring test, pulmonary function using spirometry, peripheral muscle strength using a hand-held dynamometer, muscle oxygenation using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD), static balance using the "Biosway Portable Balance System", and dynamic balance assessment using the Y balance test. The assessments will be completed in two days.

ELIGIBILITY:
Inclusion Criteria:

Cystic fibrosis patients

• Patients between the ages of 6-18 years who are diagnosed with cystic fibrosis according to the American Cystic Fibrosis Association consensus report and whose clinical condition is stable will be included in the study.

Primary ciliary dyskinesia patients • Patients between the ages of 6-18 years who are diagnosed with primary ciliary dyskinesia according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines and whose clinical condition was stable will be included in the study.

Healthy controls

• Healthy individuals of both sexes between the ages of 6-18 who voluntarily agreed to participate in the study will be included.

Exclusion Criteria:

Patients

•Patients who are uncooperative, have orthopedic or neurological disorders that will affect functional capacity, and have pneumonia or any acute infection during the evaluation will be excluded from the study.

Healthy controls;

•Those with a known chronic disease, uncooperative and orthopedic or neurological disorders that will affect functional capacity will not be included.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Thirty-one patients with CF, 27 patients with PSD were included in the study. There are 30 healthy data.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Upper extremity functional exercise capacity | First day
  Upper extremity functional exercise capacity was assessed with a 6-minute pegboard and ring test (6-PBRT). Subjects were instructed to move as many rings as possible for six minutes. Before and after each test and during the first minute of recovery, HR, SpO2, blood pressure, respiratory frequency, perceived dyspnea, and fatigue were recorded. Total ring counts were recorded as the outcome measure.

SECONDARY OUTCOMES:
Pulmonary function (Forced vital capacity (FVC)) | First day
  Pulmonary function was assesed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, forced vital capacity (FVC) was assessed.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, forced expiratory volume in the first second (FEV1) was assessed.
Pulmonary function (FEV1 / FVC) | First day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, FEV1 / FVC was assessed.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) was assessed.
Pulmonary function (Peak flow rate (PEF)) | First day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, peak flow rate (PEF) was assessed.
Peripheral muscle strength | Second day
  Quadriceps and deltoid muscle strength was assessed using a hand dynamometer (JTECH Power Track Commander, Baltimore, USA). The assessments for both the right and left sides were repeated three times.
Muscle oxygenation (SmO2rest) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (SmO2min) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (SmO2max) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (Δ SmO2) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (SmO2averaged-min) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (SmO2averaged -max) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (Δ SmO2averaged) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (SmO2recovery) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (SmO2recovery-averaged) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (THbrest) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (THbmin) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (Thbmax) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (Δ THb) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Muscle oxygenation (THbrecovery) | First day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the deltoid muscle of the dominant arm, and measurements were recorded.
Static Balance | Second day
  The static balance evaluated individuals using the "Biosway Portable Balance System" (Biodex Medical Systems Incorporated, Shirley, New York). In the evaluations, the test was repeated three times with a test duration of 20 seconds, and a 10-second inter-evaluation was permitted. The test was repeated under the conditions of eyes open, hard ground, eyes closed, hard ground, eyes open, soft ground, and eyes closed, soft ground.
Dynamic balance | Second day
  The dynamic balance assessment was evaluated using the Y balance test. The evaluations were repeated three times for both lower extremities in the anterior, posteromedial, and posterolateral directions. While the individuals maintained a single-leg stance on the right side, the left foot was extended as far as possible along the measuring tape, with the toe positioned in the anterior, posteromedial, and posterolateral directions. The same procedure was repeated on the other side.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma MUTLU KAYAARSLAN, MSc, Study Chair — Baskent University; Meral BOŞNAK GÜÇLÜ, Prof. Dr, Study Director — Gazi University; Betül YOLERİ, MSc, Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physiotherapy ana Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma R, Florea VG, Bolger AP, Doehner W, Florea ND, Coats AJ, Hodson ME, Anker SD, Henein MY. Wasting as an independent predictor of mortality in patients with cystic fibrosis. Thorax. 2001 Oct;56(10):746-50. doi: 10.1136/thorax.56.10.746. PMID 11562511
- [Background] Lucas JS, Barbato A, Collins SA, Goutaki M, Behan L, Caudri D, Dell S, Eber E, Escudier E, Hirst RA, Hogg C, Jorissen M, Latzin P, Legendre M, Leigh MW, Midulla F, Nielsen KG, Omran H, Papon JF, Pohunek P, Redfern B, Rigau D, Rindlisbacher B, Santamaria F, Shoemark A, Snijders D, Tonia T, Titieni A, Walker WT, Werner C, Bush A, Kuehni CE. European Respiratory Society guidelines for the diagnosis of primary ciliary dyskinesia. Eur Respir J. 2017 Jan 4;49(1):1601090. doi: 10.1183/13993003.01090-2016. Print 2017 Jan. PMID 27836958
- [Background] Gosselink R, Troosters T, Decramer M. Peripheral muscle weakness contributes to exercise limitation in COPD. Am J Respir Crit Care Med. 1996 Mar;153(3):976-80. doi: 10.1164/ajrccm.153.3.8630582.
- [Background] Mutlu S, Bosnak Guclu M, Sismanlar Eyuboglu T, Aslan AT. Upper Extremity Exercise Capacity and Muscle Oxygenation in Patients With Primary Ciliary Dyskinesia. Pediatr Pulmonol. 2025 Jan;60(1):e27470. doi: 10.1002/ppul.27470. PMID 39785198
- [Background] Souza RP, Donadio MVF, Heinzmann-Filho JP, Baptista RR, Pinto LA, Epifanio M, Marostica PJC. THE USE OF ULTRASONOGRAPHY TO EVALUATE MUSCLE THICKNESS AND SUBCUTANEOUS FAT IN CHILDREN AND ADOLESCENTS WITH CYSTIC FIBROSIS. Rev Paul Pediatr. 2018 Oct-Dec;36(4):457-465. doi: 10.1590/1984-0462/;2018;36;4;00015. PMID 30540111
- [Background] Halbeisen FS, Goutaki M, Spycher BD, Amirav I, Behan L, Boon M, Hogg C, Casaulta C, Crowley S, Haarman EG, Karadag B, Koerner-Rettberg C, Loebinger MR, Mazurek H, Morgan L, Nielsen KG, Omran H, Santamaria F, Schwerk N, Thouvenin G, Yiallouros P, Lucas JS, Latzin P, Kuehni CE. Lung function in patients with primary ciliary dyskinesia: an iPCD Cohort study. Eur Respir J. 2018 Aug 23;52(2):1801040. doi: 10.1183/13993003.01040-2018. Print 2018 Aug. PMID 30049738
- [Background] Harun SN, Wainwright C, Klein K, Hennig S. A systematic review of studies examining the rate of lung function decline in patients with cystic fibrosis. Paediatr Respir Rev. 2016 Sep;20:55-66. doi: 10.1016/j.prrv.2016.03.002. Epub 2016 Mar 14. PMID 27259460
- [Background] Ratjen F, Bell SC, Rowe SM, Goss CH, Quittner AL, Bush A. Cystic fibrosis. Nat Rev Dis Primers. 2015 May 14;1:15010. doi: 10.1038/nrdp.2015.10. PMID 27189798